CLINICAL TRIAL: NCT04961021
Title: Management of Consecutive Exotropia and Its Effect on Ocular Motility
Brief Title: Management of Consecutive Exotropia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Farag Khalil Ibrahiem, Assistant Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Strabismus
Record Dates: First submitted 2021-07-09; First posted 2021-07-14 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Strabismus; Concomitant Squint; Divergent Strabismus
MeSH Terms: conditions — Strabismus; Exotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medial rectus advancement with resection (Active Comparator): Surgery will be done to strengthen the medial rectus muscle with resection and anterior displacement again to the original insertion site 5 mm from limbus
  Interventions: Procedure: Strabismus surgery
- Medial rectus advancement with lateral rectus recession (Active Comparator): Surgery will be done to strengthen the medial rectus muscle with anterior displacement again to the original insertion site 4- 5 mm from limbus with weakening procedure to the lateral rectus muscle at the same time
  Interventions: Procedure: Strabismus surgery

INTERVENTIONS:
Procedure: Strabismus surgery — Strengthening of medial rectus muscle or strengthening of medial rectus muscle with weakening of the lateral rectus muscle

SUMMARY:
Patients with consecutive exotropia will be managed by medial rectus muscle advancement +/- resection or medial rectus muscle advancement +/- lateral rectus recession

ELIGIBILITY:
Inclusion Criteria:

* Patients with consecutive exotropia.
* Eight years old or more.
* Cooperative patients.

Exclusion Criteria:

* Adduction deficit.
* Mental disability.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with satisfactory postoperative alignment | 6 months
  Efficacy of each surgical procedure and its further effect using prism cover test to access postoperative alignment of the eye

CONTACTS AND LOCATIONS:
Overall Officials: Sahar TA Abdelaziz, MD, Principal Investigator — Faculty of Medicine, Minia University
Locations (1):
- Faculty of Medicine, Minya, Minya Governorate, Egypt